CLINICAL TRIAL: NCT03439579
Title: Pilot Study of the Home Weight Loss Program
Brief Title: Pilot Study of the HWL Program
Acronym: HWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: South Carolina Telehealth Alliance (Other)
Responsible Party: Principal Investigator, Patrick O'Neil, Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00070941
Record Dates: First submitted 2018-02-07; First posted 2018-02-20 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Overweight and Obesity
Keywords: Telehealth; Remote weight loss; Self-monitoring; Diet; Physical activity
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single group pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home weight loss program (Experimental): Participants will be instructed to daily monitor their body weight, minutes of activity, number of steps, and calories consumed for the duration of the pilot study, and they will receive recorded individualized feedback on this self-monitored data from Weight Management Center clinicians (registered dietitians, exercise psychologists, and behavioral specialists).
  Interventions: Behavioral: Home weight loss program

INTERVENTIONS:
Behavioral: Home weight loss program — Patient remote self-monitoring of diet, activity, and weight with clinician feedback provided remotely based on self-monitored data.

SUMMARY:
The goal of the project is to test a remotely delivered, standalone behavioral weight loss intervention designed to help adults initiate the important dietary, physical activity (PA) and behavioral changes necessary to achieve weight loss.

DETAILED DESCRIPTION:
The Weight Management Center currently offers a remotely delivered (smart phone, tablet, computer) program to assist patients with maintaining weight losses already achieved, which includes multi-channel self-monitoring and asynchronous individually recorded feedback from clinical staff. The goal of the presently proposed project is to build on this existing maintenance-focused program to create a remotely delivered, standalone behavioral weight loss intervention designed to help participants initiate the important dietary, physical activity (PA) and behavioral changes necessary to achieve weight loss. We recently developed the Home Weight Loss (HWL) program by repackaging existing clinical educational materials as instructional lifestyle change modules to be delivered remotely for participant weight loss

The aim of the proposed project are to pilot test the effects of the HWL program among a sample of overweight and obese adults (N=30). The digital platform currently used in the maintenance program will be used for the HWL program

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years
* BMI = 25.0- 40 kg/m2
* Internet access via desktop or laptop computer
* valid email address
* smart phone ownership
* women of childbearing potential must agree to use effective contraception during the study

Exclusion Criteria:

* currently dieting (>10-pound weight loss in past 3 months)
* another member of the household is participating in this pilot study
* inability to engage in physical activity
* inability to read and speak English
* diagnosis of diabetes (other than treated by diet alone),
* uncontrolled thyroid condition or other endocrine disorder
* major depressive disorder or other severe psychiatric disorder (e.g., bipolar disorder) within the past two years
* past suicide attempt
* current use of prescription or over-the-counter weight loss medications
* current/planned pregnancy
* drug and/or alcohol abuse
* use of steroid medication for more than 10 days in the past three months *implanted electronic devices

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Body weight change | 12 weeks
  body weight change (kg) from pre-to post

SECONDARY OUTCOMES:
changes in body weight as a percentage of start weight | 12 weeks
  percent body weight change
changes in body mass index | 12 weeks
  weight in kgs divided by height in meters squared to obtain BMI (kg/m^2)
program satisfaction | 12 weeks
  program satisfaction obtained from multiple choice items developed by study staff. Subjects are asked to rate their level of agreement with items assessing their satisfaction with the overall program, available responses range from extremely satisfied to not at all satisfied.
changes in body fat percentage | 12 weeks
  changes in body fat percentage
changes in waist and hip measurements | 12 weeks
  changes in waist and hip measurements
usability of program components | 12 weeks
  examine usage of tracking components including step, exercise, diet, and weight tracking
changes in eating behavior scores | 12 weeks
  use of the Eating Behavior Inventory (EBI). This is a validated 26-item scale assessing eating and weight control behaviors. Subjects indicate agreement with statements with reponse options ranging in values from 1 (never or hardly ever) to 5 (always or almost). Higher values are indicative of those most associated with weight loss (e.g., self-monitoring caloric intake) and are therefore associated with better weight loss outcomes following behavioral weight management intervention.
changes in scores on the power of food scale | 12 weeks
  use of the Power of Food Scale (PFS). This is a validated 15-item scale with responses scored and ranging between 1 (do not agree) and 5 (strongly agree) with the statements. Higher scores indicate less favorable outcomes, as higher scores indicate increased patient susceptibility to food in the environment.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M O'Neil, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No individual data is planned to be shared with other researchers.